CLINICAL TRIAL: NCT06454370
Title: Histopathological Analysis of Minor Salivary Gland Biopsy Following Dynamic Full-field Optical Coherence Tomography, a Comparison to Conventional Histopathological Findings in Patients Suspect Sjogren Syndrome.
Brief Title: Histopathological Analysis Versus Full-field Optical Coherence Tomography of Minor Salivary Gland Biopsy in Suspect Sjogren Syndrome
Acronym: TOCOSS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Mâcon (Other)
Collaborators: Centre Hospitalier William Morey - Chalon sur Saône (Other); Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: TOCOSS
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Sjogren's Syndrome; Tomography Optical Coherence
Keywords: Minor Salivary gland biopsy; Tomography, Optical Coherence
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary Sjögren syndrome (pSS) is a systemic autoimmune disease that mainly affects the exocrine glands leading to severe dryness of mucosal surfaces, principally in the mouth and eyes. The other clinical manifestations are fatigue and musculoskeletal pain. Diagnosis of pSS associates clinical abnormalities with specific antibodies (Ro/SSA and La/SSB antibodies) or histopathological criteria of a minor salivary gland biopsy (the presence and number of lymphocytic focus, as well as chronicity findings like acinar atrophy, ductal dilatation or fibrosis). Apart from its variable sensitivity, one of the weaknesses of minor salivary gland biopsy is the delay in obtaining the result due to the time required to prepare the sample for histological analysis.

Our group recently demonstrated the use of full-field optical coherence tomography (FF-OCT) to visualize structural changes associated with the inflammatory processes in Giant Cell Arteritis (temporal artery biopsy examination). It may suggests a further use of dynamic FF-OCT of minor salivary gland biopsy to visualize structural changes associated with the lymhocytic focus to ensure rapid on-site diagnosis of pSS.

DETAILED DESCRIPTION:
This study does not require additional examination, and will use the data performed from the minor salivary gland biopsy carried out as part of usual care, in comparison with the results of the conventional histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years of age with suspected Sjogren Syndrome received minor gland salivary biopsy

Exclusion Criteria:

* Inability to perform dynamic full-field optical coherence tomography observation at the moment of temporal artery biopsy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TOCOSS cohort : Patient > 18 years old with suspected Sjogren Syndrome received minor gland salivary biopsy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-10-07 (Estimated); Study Completion 2024-12-07 (Estimated)

PRIMARY OUTCOMES:
Histopathological analysis of healthy minor salivary gland biopsy with dynamic full-field optical coherence tomography | Outcome measure is assessed 15 days following minor salivary gland biopsy
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify the normal structures of a minor salivary gland biopsy, i.e . salivary parenchyma with secretory units arranged into acini (group of acinar cells organized around a narrow lumen)

SECONDARY OUTCOMES:
Histopathological analysis of Sjogren's syndrom minor salivary gland biopsy with dynamic full-field optical coherence tomography | Outcome measure is assessed 15 days following minor salivary gland biopsy
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify histopathological features of Sjogren syndrom, i.e. lymphocytic foci, particularly located in the periductal area (according to the classification defined by Chisholm and Mason), acinar atrophy, ductal dilatation, and fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Thibault MAILLET, Principal Investigator — Internal Medicine - Centre Hospitalier de Mâcon
Locations (1):
- Centre Hospitalier de Mâcon, Mâcon, Sâone-et-Loire, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manuel RC, Pilar BZ, Raphaele S, Hendrika B, Simon J B, Thomas D, Jacques-Eric G, Xavier M, Elke T, Stefano B, Salvatore V, Thomas M, Wan-Fai N, Aike K, Athanasios T, Claudio V; EULAR Sjogren Syndrome Task Force. Characterization of systemic disease in primary Sjogren's syndrome: EULAR-SS Task Force recommendations for articular, cutaneous, pulmonary and renal involvements. Rheumatology (Oxford). 2017 Jul 1;56(7):1245. doi: 10.1093/rheumatology/kex157. No abstract available. PMID 28379527
- [Result] Shiboski CH, Shiboski SC, Seror R, Criswell LA, Labetoulle M, Lietman TM, Rasmussen A, Scofield H, Vitali C, Bowman SJ, Mariette X; International Sjogren's Syndrome Criteria Working Group. 2016 American College of Rheumatology/European League Against Rheumatism Classification Criteria for Primary Sjogren's Syndrome: A Consensus and Data-Driven Methodology Involving Three International Patient Cohorts. Arthritis Rheumatol. 2017 Jan;69(1):35-45. doi: 10.1002/art.39859. Epub 2016 Oct 26. PMID 27785888
- [Result] Maldiney T, Greigert H, Martin L, Benoit E, Creuzot-Garcher C, Gabrielle PH, Chassot JM, Boccara C, Balvay D, Tavitian B, Clement O, Audia S, Bonnotte B, Samson M. Full-field optical coherence tomography for the diagnosis of giant cell arteritis. PLoS One. 2020 Aug 31;15(8):e0234165. doi: 10.1371/journal.pone.0234165. eCollection 2020. PMID 32866179